CLINICAL TRIAL: NCT01720173
Title: A Phase II Evaluation of Dalantercept (NSC #757172), a Novel Soluble Recombinant Activin Receptor-Like Kinase 1 (ALK-1) Inhibitor Receptor-Fusion Protein, in the Treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Brief Title: Dalantercept in Treating Patients With Recurrent Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0170R; NCI-2012-01936 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NSC #757172; CDR0000742512; GOG-0170R (Other: NRG Oncology); GOG-0170R (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2012-10-30; First posted 2012-11-02 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — ALK1-Fc fusion protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dalantercept) (Experimental): Patients receive dalantercept SC on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dalantercept; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Dalantercept — Given SC
  Other Names: ACE-041; Activin Receptor-like Kinase 1 Inhibitor ACE-041; ALK1-Fc Fusion Protein ACE-041
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well dalantercept works in treating patients with ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer that has returned. Dalantercept may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Dalantercept may also stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients who survive progression-free for at least 6 months and the proportion of patients who have objective tumor response (complete or partial) in patients with persistent or recurrent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma, treated with dalantercept.

II. To determine the frequency and severity of adverse events associated with treatment with dalantercept as assessed by the Active Version of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OBJECTIVES:

I. To determine the duration of progression-free survival (PFS) and overall survival (OS).

TERTIARY OBJECTIVES:

I. To measure the expression of vascular endothelial growth factor (VEGF), fibroblast growth factor (FGF), platelet-derived growth factor (PDGF), transforming growth factor-beta (TGF-B), activin receptor-like kinase 1 (ALK1), cluster of differentiation 105 (CD105), and other markers via immunohistochemistry (IHC) and determine if there is correlation between expression and clinical response to treatment.

II. To determine the correlation between ALK1 gene expression, other markers, and clinical response to treatment.

III. To determine the correlation between concentration of VEGF, bone morphogenetic protein (BMP)9, BMP10, and ALK1 in pre-cycle 1 plasma using an enzyme-linked immunosorbent assay (ELISA), and clinical response to treatment.

OUTLINE:

Patients receive dalantercept subcutaneously (SC) on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma; histologic documentation of the original primary tumor is required via the pathology report
* All patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patient must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase III protocol or Rare Tumor protocol for the same patient population
* Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2; patients who have received two prior regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy:

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted
  * Any other prior therapy directed at the malignant tumor, including immunologic agents, must be discontinued at least three weeks prior to registration; therapy with nitrosoureas or mitomycin must be discontinued at least six weeks prior to registration
  * Any prior radiation therapy must be discontinued at least four weeks prior to registration
  * At least 4 weeks must have elapsed since the patient underwent any major surgery (e.g., major: laparotomy, laparoscopy); there is no delay in treatment for minor procedures (e.g., central venous access catheter placement)
* Prior therapy:

  * Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, consolidation, biologic/targeted (non-cytotoxic) agents (e.g., bevacizumab) or extended therapy administered after surgical or non-surgical assessment
  * Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease
  * Patients who have received only one prior cytotoxic regimen (platinum-based regimen for management of primary disease), must have a platinum-free interval of less than 12 months, or have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
  * Patients are allowed to receive, but are not required to receive, biologic/targeted (non-cytotoxic) therapy as part of their primary treatment regimen
  * Patients must have NOT received any biologic/targeted (non-cytotoxic) therapy targeting the VEGF pathway for management of recurrent or persistent disease
  * For the purposes of this study, poly (ADP-ribose) polymerase (PARP) inhibitors will be considered ?cytotoxic?; patients are allowed to receive, but are not required to receive, PARP inhibitors for management of primary or recurrent/persistent disease (either alone or in combination with cytotoxic chemotherapy); PARP inhibitors will NOT count as a prior regimen when given alone
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to100,000/mcl
* Hemoglobin greater than or equal to 9 g/dl
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN)
* Sodium greater than or equal to 130 mEq/L (CTCAE version 4 [v. 4], grade 0 or 1)
* Urine protein should be screened by urinalysis; if protein is 2+ or higher, 24-hour urine protein should be obtained and the level should be < 1000 mg (< 1.0 g/24 hrs) for patient enrollment
* Bilirubin less than or equal to 1.5 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 3 x ULN
* Albumin greater than or equal to 3 (CTCAE v. 4, grade 0 or 1)
* Prothrombin time (PT) such that international normalized ratio (INR) is less than or equal to 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and partial thromboplastin time (PTT) less than or equal to 1.5 x ULN
* Left ventricular ejection fraction (LVEF) greater than 50% (measured by echocardiogram or MUGA [multi-gated acquisition] scan)
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements
* Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception

Exclusion Criteria:

* Patients who have had previous treatment with dalantercept or any other anti-ALK1 (activin receptor-like kinase 1) agent
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with a past history of primary endometrial cancer are excluded unless all of the following conditions are met: stage not greater than I-B; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serious, clear cell or other International Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions
* Patients with history or evidence upon physical exam of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy or any brain metastases
* Serious or non-healing wound, ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months
* Patients requiring parenteral hydration or parenteral/total parenteral nutrition
* Patients with:

  * Active bleeding (e.g., active hemoptysis, defined as bright red blood of greater than or equal to 1/2 teaspoon [2.5 ml] in any 24 hour period within 2 weeks prior to registration or gastrointestinal bleeding within 3 months prior to registration)
  * Hereditary hemorrhagic telangiectasia (HHT)
  * Platelet function abnormality
  * Autoimmune or hereditary hemolysis
  * Coagulopathy
  * Tumor involving major vessels (defined as any lesion invading or abutting the wall [i.e., no fat plane evident] of major blood vessels as assessed by CT or MRI)
* Patients receiving treatment with full dose aspirin (325mg oral daily), clopidogrel (Plavix) or dabigatran (Pradaxa)
* Patients with peripheral edema greater than or equal to grade 1, within 4 weeks of registration
* Patients with clinically significant cardiovascular disease:

  * Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg despite antihypertensive medications
  * Evidence of hypertrophic cardiomyopathy
  * New York Heart Association (NYHA) class II or greater congestive heart failure (CHF)
  * Any of the following within 6 months prior to study registration:

    * Bypass surgery
    * Stent placement
    * Myocardial infarction
    * Acute coronary syndrome/unstable angina
    * Hospitalization for CHF
  * Serious cardiac arrhythmia requiring medication; this does not include asymptomatic, atrial fibrillation with controlled ventricular rate
  * Prolonged corrected QT (QTc) interval > 450 ms
  * Prior anthracycline cumulative dose > 450 mg/m^2
* History of severe (National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] v.4.0 >= grade 3) allergic or anaphylactic reaction or hypersensitivity to recombinant proteins or Tris buffered saline
* Patients who are pregnant or nursing
* History of syndrome of inappropriate antidiuretic hormone secretion (SIADH)
* Patients who have undergone a therapeutic paracentesis within 4 weeks of registration
* Known history of positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody, or human immunodeficiency virus (HIV) antibody results
* Clinically significant active pulmonary risk including pulmonary hypertension, pulmonary embolism, or history of pulmonary edema

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11-05 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Burger, Principal Investigator — NRG Oncology
Locations (40):
- United States (40):
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Decatur Memorial Hospital, Decatur, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Christiana Care - Union Hospital, Elkton, Maryland
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford NCI Community Oncology Research Program of the North Central Plains, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Pacific Gynecology Specialists, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 11/5/2012 and closed to accrual on 10/2/2013.
Groups:
- Dalantercept: Dalantercept administered subcutaneously at a dose of 1.2mg/kg (maximum starting dose of 120 mg*) once every three weeks until disease progression or adverse effects prohibit further therapy. One cycle is 3 weeks.
  *Patients weighing more than 100kg will start treatment at 120mg, and if dalantercept is tolerated for 2 cycles (i.e. toxicities are tolerable, less than grade 2 and resolved), the patient can be dose escalated to dosing based on actual body weight.
Period: Overall Study
Arm/Group | Dalantercept
Started | 30
Completed (Eligible and treated patients.) | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Dalantercept
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (9.2)
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 1
  40-49 years | 6
  50-59 years | 13
  60-69 years | 5
  70-79 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free for at Least 6 Months Without Non-protocol Therapy From Study Entry
Description: Percentage of participants who survive progression-free for at least 6 months without non-protocol therapy after study entry. Progression is assessed by RECIST 1.1. RECIST 1.1 defines progressive disease as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions or unequivocal progression of non-target lesions is also considered progression.
Time Frame: Every other cycle for first 6 months
Population: Eligible and treated participants
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dalantercept
Number analyzed (Participants) | 30
percentage of participants | 20 [11 to 100]

2. Primary Outcome: Incidence of Adverse Effects as Assessed by Common Terminology Criteria for Adverse Events Version 4.0
Description: Number of participants with a maximum grade of 3 or higher during the treatment period.
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Dalantercept
Number analyzed (Participants) | 30
Participants
  Neutropenia | 1
  Other Investigations | 1
  Cardiac disorders | 3
  Gastrointestinal disorders | 2
  General disorders and administration site conditio | 2
  Infections and infestations | 3
  Metabolism and nutrition disorders | 1
  Musculoskeletal and connective tissue disorders | 1
  Renal and urinary disorders | 1
  Reproductive system and breast disorders | 1
  Respiratory, thoracic and mediastinal disorders | 1

3. Primary Outcome: Objective Tumor Response
Description: Complete and Partial Tumor Response by RECIST 1.1. RECIST 1.1 defines complete response as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and the disappearance of all non-target lesions and normalization of tumor marker level. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: Every other cycle for first 6 months; then every 3 months thereafter until disease progression confirmed; and at any other time if clinically indicated based on symptoms or physical signs suggestive of progressive disease, up to 5 years.
Population: Eligible and treated participants
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dalantercept
Number analyzed (Participants) | 30
percentage of participants | 0 [0 to 100]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years.
Population: Eligible and treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dalantercept
Number analyzed (Participants) | 30
months | 19.8 [8.8 to 24.4]

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is the period of time from study entry to time of disease progression, death or date of last contact, whichever occurs first. Progression is assessed by RECIST 1.1. RECIST 1.1 defines progressive disease as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions or unequivocal progression of non-target lesions is also considered progression.
Time Frame: as for outcome 3
Population: Eligible and treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dalantercept
Number analyzed (Participants) | 30
months | 1.7 [1.3 to 3.7]

6. Other Pre Specified Outcome: Gene Expression Levels of ALK1 and Other Markers
Description: Associated with measures of clinical response to treatment, including PFS and OS.
Time Frame: Baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: IHC Expression Levels of VEGF, FGF, TGFB, ALK1, CD105 and Other Markers
Description: Associated with measures of clinical response to treatment, including PFS and OS.
Time Frame: Baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Pre-treatment Plasma Concentration Levels of VEGF, BMP9, BMP10, and ALK1
Description: Associated with measures of clinical response to treatment, including PFS and OS.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. The average time of study treatment was 3 months.
Arm/Group | Dalantercept
Serious Adverse Events (participants affected / at risk) | 8/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalantercept (N=30)
Colonic Obstruction (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Dysphasia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalantercept (N=30)
Lymph Node Pain (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 21
Palpitations (Cardiac disorders) | 3
Heart Failure (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Ear Pain (Ear and labyrinth disorders) | 2
Hyperparathyroidism (Endocrine disorders) | 1
Eye Disorders - Other (Eye disorders) | 1
Blurred Vision (Eye disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 6
Bloating (Gastrointestinal disorders) | 4
Abdominal Pain (Gastrointestinal disorders) | 14
Oral Dysesthesia (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 1
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1
Oral Hemorrhage (Gastrointestinal disorders) | 2
Oral Pain (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 8
Fecal Incontinence (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 6
Flatulence (Gastrointestinal disorders) | 1
Pain (General disorders) | 2
Malaise (General disorders) | 2
Localized Edema (General disorders) | 1
Injection Site Reaction (General disorders) | 1
Edema Trunk (General disorders) | 2
Non-Cardiac Chest Pain (General disorders) | 1
Edema Limbs (General disorders) | 11
Edema Face (General disorders) | 1
Fatigue (General disorders) | 20
Fever (General disorders) | 5
Chills (General disorders) | 3
Allergic Reaction (Immune system disorders) | 1
Peripheral Nerve Infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Lip Infection (Infections and infestations) | 1
Weight Loss (Investigations) | 1
Weight Gain (Investigations) | 8
Platelet Count Decreased (Investigations) | 6
Lymphocyte Count Decreased (Investigations) | 1
Creatinine Increased (Investigations) | 3
Neutrophil Count Decreased (Investigations) | 2
White Blood Cell Decreased (Investigations) | 6
Aspartate Aminotransferase Increased (Investigations) | 3
Alkaline Phosphatase Increased (Investigations) | 3
Alanine Aminotransferase Increased (Investigations) | 3
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Peripheral Sensory Neuropathy (Nervous system disorders) | 10
Peripheral Motor Neuropathy (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 3
Memory Impairment (Nervous system disorders) | 1
Headache (Nervous system disorders) | 15
Dizziness (Nervous system disorders) | 3
Cognitive Disturbance (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 1
Urinary Tract Pain (Renal and urinary disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 1
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Periorbital Edema (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5
Telangiectasia (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Thromboembolic Event (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less